CLINICAL TRIAL: NCT05471583
Title: Assessment of Endothelial Glycocalyx Dysfunction and Impaired Microcirculatory Perfusion During Cardiac Surgery to Improve Prediction of Post-operative Acute Kidney
Brief Title: Endothelial Glycocalyx Damage in Acute Kidney Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: King's College Hospital NHS Trust (Other); British Heart Foundation (Other)
Responsible Party: Principal Investigator, Dr Jennifer Joslin, Clinical Research Fellow, King's College London
Other Study IDs: KCH19-107
Record Dates: First submitted 2022-03-30; First posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Coronary Artery Disease; Acute Kidney Injury
Keywords: endothelial glycocalyx; microvascular perfusion
MeSH Terms: conditions — Coronary Artery Disease; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma, serum, (spun urine)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Main group: There is only one group in the study. It is observational.
  Interventions: Other: Main group

INTERVENTIONS:
Other: Main group — no intervention; observational only

SUMMARY:
Abstract Significance: Cardiac surgery-associated acute kidney injury (CSA-AKI) is common and has serious immediate and long-term sequelae. Better early prediction of those at highest risk and greater understanding of underlying pathological processes are needed to prevent or minimise damage.

Hypotheses

* Dynamic changes in systemic endothelial glycocalyx (Glx) and microcirculatory parameters during coronary artery bypass graft (CABG) surgery are predictive of CSA-AKI.
* Mechanisms for Glx degradation during CABG surgery are akin to those during sepsis Aims
* Investigate Glx and microcirculatory health throughout CABG surgery and recovery and their association with CSA-AKI.
* Explore association between inflammation and Glx degradation during CABG surgery.

Methodology

1. Prospective cohort study: serial sampling and microcirculatory perfusion imaging of 70 patients undergoing CABG surgery with evaluation of CSA-AKI predictors, including plasma Syndecan-1.
2. Examination of inflammation and cardiometabolic proteome and association with vascular changes
3. In vitro mechanistic assessment of Glx degradation and relative timing of organelle exocytosis in cultured endothelial cells in response to patient serum, targeting identified candidate mediators.

Impact: Enhancing CSA-AKI risk stratification with new mechanistic biomarkers will enable individualised management of at-risk patients, and pathophysiological insights will create possible therapeutic targets, thus reducing morbidity, mortality and cost of CSA-AKI.

DETAILED DESCRIPTION:
Study design: Prospective cohort study.

The investigators will recruit 70 elective patients undergoing CABG surgery with and without cardiopulmonary bypass (CPB), with blood and urine sampling and assessment of microcirculatory perfusion by IDF in pre- peri- and post-operative periods, with informed written consent. The investigators have completed a feasibility study with successful recruitment and data collection at all time points and the current protocol and patient material have been reviewed by a patient representative.

Blood and urine samples will be analysed to consider markers of endothelial glycocalyx degradation (including syndecan-1 (SDC1)), endothelial activation (including thrombomodulin (TM)), and markers of renal tubular stress (NephroCheck).

Sublingual microcirculatory perfusion assessed by IDF imaging is painless and low risk and participant acceptability has been confirmed during the feasibility study. The process involves using a small handheld probe to gently press on the underside of the tongue and takes 3-10 minutes. Four video clips of 10s will be taken from each participant from different sites within the sublingual area. Videos will be exported as pseudonymised files for analysis. Image collection and analysis will be performed in accordance with international consensus recommendations, using a CytoCam video-microscope (Braedius Medical B.V., Huizen, The Netherlands). Images will be analysed using a dedicated software tool (Automated Vascular Analysis V.3.02, Microvision Medical, The Netherlands). Data generated will include flow and density-based measures of the microcirculation, including Perfused Vessel Density (PVD) and Microcirculatory Flow Index (MFI).

Peri-operative sampling and imaging will occur at predefined surgical time-points, in keeping with previous studies and informed by the feasibility study. Time-points were selected in anticipation of the most informative results, including point of peak "reperfusion" after final surgical anastomosis, and to minimise participant inconvenience (existing arterial line and urinary catheter tubing will be used) and to avoid surgical disruption and delays (IDF is quicker during anaesthesia and previous studies have shown negligible change between baseline and assessment immediately after anaesthesia prior to surgery).

Confounding factors: Factors affecting development of AKI include medical history (chronic kidney disease, hypertension, diabetes), surgical factors (operation, CPB and aortic cross clamp duration, use of blood products), free haemoglobin (fHb) and macrovascular parameters (blood pressure, lactate, cardiac output, haematocrit) will be recorded and statistical analyses adjustment performed.

Follow up: Until seven days post-op or discharge from hospital, whichever is soonest.

Proposed sample size: 70 (single centre study)

Power calculations: The cohort study is powered to determine the primary outcome: peak plasma SDC1 concentration between those who do and do not develop CSA-AKI. The investigators' retrospective analysis found post-CABG CSA-AKI incidence in their hospital to be 19%. The most appropriate published study offering test statistics to guide the power calculation is one of AKI in a cohort of patients with acute decompensated heart failure. The difference in mean SDC1 between those with and without AKI (effect size) was calculated from presented data as 153.2±123.8ng/ml. Assuming a power value of 80% and significance level of 5%, a calculation using the T statistic yields a sample of 36: 7 with CSA-AKI and 29 without. The investigators have further repeated the calculations using unpublished data from patients with traumatic haemorrhagic shock, where the difference in mean SDC1 between those with and without AKI was 175.2±185.5ng/ml. With the same assumptions as previously, the calculation yields a sample of 61: 12 with CSA-AKI and 49 without. The investigators will use the more conservative of these calculations, allow for a 10% dropout rate, and aim to recruit 70 patients.

Loss to follow-up: As all sampling and data collection will take place over a very short period there should be no loss to follow-up, as in the feasibility study. If participants withdraw consent then no further samples or images will be collected.

Bias: Participants will be recruited by consecutive convenience sampling. There is unlikely to be any differences between those approached and not approached, and selection bias is unlikely to apply. Information bias is also unlikely as all measurements and data to be collected is objective. The investigators will protect against assessment bias when analyzing results by pseudonymisation of samples and IDF videos. Confounding factors will be accounted for during analysis, as above.

Statistical analysis: Patients will be divided into two groups based on CSA-AKI presence or absence. The difference between peak SDC1 between groups will be assessed using T-tests. Multiple logistic regression with AKI as the outcome and peak SDC1 as independent predictor will be used to consider confounding parameters, including fHb. P-values <0.05 will be considered statistically significant. Analysis will be repeated for difference between peak SDC1 and baseline for each participant, to take into account possible pre-existing glycocalyceal injury. Correlation between SDC1 and TM and PVD / MFI will be calculated, using either continuous variables or categorical groups as appropriate. To determine the predictive value of SDC1 and microcirculatory variables in CSA-AKI receiver operating characteristic (ROC) curves will be constructed for each variable by plotting sensitivity versus (1-specificity) for a series of threshold values and calculating the area under the curve (AUC) for each. These will be compared to those for NephroCheck score, Cleveland Clinic Score, fHb, lactate, and macrovascular parameters.

Data access: Data collected during this study will only be accessible to the study team, and to the Sponsor for regulatory purposes.

Data and sample storage: All data will be stored in accordance with Caldicott Principles.

ELIGIBILITY:
Inclusion Criteria:

* Listed for CABG surgery with or without CPB, age >18 years, able and willing to give written informed consent.

Exclusion Criteria:

* Unable / unwilling to provide blood samples or undergo IDF imaging, cross-clamp fibrillation technique, already on renal replacement therapy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults scheduled to undergo CABG at King's College Hospital (KCH)
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-11-16 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Acute kidney injury | 7 days
  as per Kidney Disease Improving Global Outcomes (KDIGO) guidelines

SECONDARY OUTCOMES:
thrombomodulin change | through study completion: 24 hours
  change in concentration of plasma thrombomodulin between groups with and without AKI
NephroCheck | 1 hour post-op
  urinary NephroCheck between groups with and without AKI
Syndecan-1 change | through study completion: 24 hours
  change in concentration of plasma syndecan-1 between groups with and without AKI
microvascular flow index | up to 1 hour post-op
  microvascular flow index between groups with and without AKI
perfused vessel density | up to 1 hour post-op
  perfused vessel density between groups with and without AKI

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No